CLINICAL TRIAL: NCT00330330
Title: A Double-Blind, Placebo-Controlled, Dose-Escalation Study to Assess the Safety, Tolerability, Pharmacokinetics, and Activity of ISIS 113715 in Patients With Type 2 Diabetes Mellitus Who Have Not Received Prior Therapy
Brief Title: Safety, Tolerability, and Activity of ISIS 113715 in People With Type 2 Diabetes Mellitus Who Have Not Received Prior Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ISIS 113715-CS7
Record Dates: First submitted 2006-05-24; First posted 2006-05-26 (Estimated); Last update posted 2008-02-06 (Estimated); Status verified 2008-02

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Fasting plasma glucose; HbA1c
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — ISIS-113715

INTERVENTIONS:
Drug: ISIS 113715

SUMMARY:
The aim of this study is to evaluate the safety, tolerability, and pharmacokinetics of five ISIS 113715 intravenous dose cohorts in drug-naïve type 2 diabetics.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes Mellitus of less than 5 years in duration
* Have never received hypoglycemic therapy
* Aged 18 to 65 years
* Fasting blood glucose between 130 and 220 mg/dL (7.2 to 12.2 mmol/L) for Cohorts A-D and between 140 and 220 mg/dL (7.8 to 12.2 mmol/L) for Cohort E
* HbA1c between 6.8 and 10.0% for Cohorts A-D and between 7.5 and 11.0% for Cohort E
* Body Mass index > 25 and < 35 kg m -2

Exclusion Criteria:

* Medication that may affect glucose homeostasis (e.g. systemic glucocorticoid) within one month of screening
* Clinically significant abnormalities in medical history or physical exam
* Clinically significant abnormalities on laboratory examination
* History of HIV infection
* Active infection requiring antiviral or antimicrobial therapy
* Malignancy (with the exception of basal or squamous cell carcinoma of the skin if adequately treated and no recurrence for > one year at the time of screening)
* Any other concurrent condition which, in the opinion of the Investigator, would preclude participation in or interfere with compliance
* Alcohol or drug abuse
* Undergoing or have undergone treatment with another investigational drug, biologic agent or device within 90 days of screening
* Abnormal serum creatinine concentration defined as > 1.5 mg/dL (132.6 micro mol/L) for males and > 1.2 mg/dL (106 micro mol/L) for females
* Medications that may affect coagulation (heparin, warfarin, etc.) with the exception of acetylsalicylic acid or non-steroidal anti-inflammatory agents.
* Allergy to sulfur-containing medications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96
Dates: Start 2003-02; Study Completion 2006-08

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of ISIS 113715
To evaluate the pharmacokinetic profile of ISIS 113715
To evaluate the pharmacologic activity of ISIS 113715

CONTACTS AND LOCATIONS:
Overall Officials: Mark K Wedel, MD, JD, FACP, Study Director — Ionis Pharmaceuticals, Inc.
Locations (10):
- Poland (3):
  - NZOZ Specjalistyczny Osrodek Internistyczno Diabetologiczny, Bialystok
  - Prywatna Praktyka Lekarska, Radom
  - Oddzial Chorob Wewnetrznych ze Stacja Dializ Szpital w Wolominie, Wołomin
- Russia (7):
  - Chair of Endocrinology and Diabetology of the Faculty of Advenced Training for Physicians, Moscow
  - Endocrinology Scientific Centre of RAMS, Moscow
  - Medical Institution "Polyclinic OAOA Gazprom", Moscow
  - Close Corporation "MEDSI", Moscow
  - Chair of Endocrinology and Diabetology Central Clinical Hospital of the Ministry of Communications of RF, Moscow
  - Moscow Regional Scientific-Research Clinical Institute named after I.F. Vladimirsky, Moscow
  - Clinic of Therapy of Postgraduate Education named after N.S. Molchanov, Saint Petersburg

REFERENCES:
- [Derived] Burel SA, Machemer T, Baker BF, Kwoh TJ, Paz S, Younis H, Henry SP. Early-Stage Identification and Avoidance of Antisense Oligonucleotides Causing Species-Specific Inflammatory Responses in Human Volunteer Peripheral Blood Mononuclear Cells. Nucleic Acid Ther. 2022 Dec;32(6):457-472. doi: 10.1089/nat.2022.0033. Epub 2022 Aug 17. PMID 35976085